CLINICAL TRIAL: NCT00086658
Title: A Multicenter, Double-blind, Placebo-controlled, Study to to Evaluate the Corticosteroid- Sparing Effects of Mepolizumab in Subjects With Hypereosinophilic Syndromes (HES) and Evaluate Efficacy and Safety of Mepolizumab in Controlling the Clinical Signs and Symptoms of Subjects With HES
Brief Title: Intravenous Mepolizumab In Subjects With Hypereosinophilic Syndromes (HES)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100185; NCT00081445 (obsolete NCT alias)
Record Dates: First submitted 2004-07-07; First posted 2004-07-09 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Hypereosinophilia; Hypereosinophilic Syndrome
Keywords: Hypereosinophilic Syndrome Hypereosinophilia; mepolizumab; anti IL-5
MeSH Terms: conditions — Eosinophilia; Hypereosinophilic Syndrome | interventions — mepolizumab

INTERVENTIONS:
Drug: mepolizumab

SUMMARY:
Hypereosinophilic syndrome (HES) is a rare disease with broad clinical signs and symptoms which is diagnosed based on a persistent blood eosinophil count of greater than 1500 cells, various end-organ damages (including skin, heart, lung, nervous system and digestive system etc.), and with exclusion of known secondary causes of hypereosinophilia.

HES has a high morbidity/mortality rate. The major treatment of HES has been systemic corticosteroid and other chemotherapeutic drugs (for example, hydroxyurea and interferon) with the intention to lower eosinophil counts and therefore to slow down the progression of disease. Even though corticosteroid and other therapies can effectively reduce eosinophilia in some patients, some may eventually become nonresponsive and intolerable to the amount of side effects of the long-term therapy with these medications.

Mepolizumab is a humanized monoclonal antibody that binds specifically to human interleukin 5 (hIL-5) and inhibits its activity. Previous human experience has shown it has been effective in reducing blood eosinophilia in atopic and HES patients and has alleviated some HES clinical signs and symptoms. This study intends to further evaluate the corticosteroid-sparing and clinical benefit of mepolizumab in HES.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Phase III Study to Evaluate Corticosteroid-reduction and -sparing effects of Mepolizumab 750 mg intravenously in Subjects with Hypereosinophilic Syndromes (HES) and to evaluate the Efficacy and Safety of Mepolizumab in controlling the Clinical Signs and Symptoms of HES over Nine Months

ELIGIBILITY:
Inclusion criteria:

* Documented history of Hypereosinophilic Syndrome (HES)
* Eosinophil count greater than 1500 cells for 6 months
* Signs and symptoms of organ system involvement
* No evidence of parasitic, allergic or other causes of eosinophilia after comprehensive evaluation.
* Achieve and maintain a stable prednisone (corticosteroid) dose prior to starting study medication.
* Not pregnant or nursing.

Exclusion criteria:

* Churg-Strauss Syndrome
* Wegener's Granulomatosis
* Lymphoma, hematological malignancy, advanced and metastatic solid tumors
* Chemotherapy, radiotherapy or interleukin 2 treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-03-23 (Actual); Primary Completion 2006-05-01 (Actual); Study Completion 2006-05-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a total daily prednisone dose of </=10 mg for a period of 8 consecutive weeks

SECONDARY OUTCOMES:
Assess the effect of mepo in lowering prednisone dose and blood eosinophil count, improving HES-associated skin manifestations, improving quality of life (QoL), safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (29):
- United States (11):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Madison, Wisconsin
- Australia (4):
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, West Perth, Western Australia
- GSK Investigational Site, Leuven, Belgium
- Canada (6):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (2):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Suresnes
- Germany (3):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bad Bramstedt, Schleswig-Holstein
- GSK Investigational Site, Bologna, Emilia-Romagna, Italy
- GSK Investigational Site, Bern, Switzerland

REFERENCES:
- [Derived] Roufosse F, de Lavareille A, Schandene L, Cogan E, Georgelas A, Wagner L, Xi L, Raffeld M, Goldman M, Gleich GJ, Klion A. Mepolizumab as a corticosteroid-sparing agent in lymphocytic variant hypereosinophilic syndrome. J Allergy Clin Immunol. 2010 Oct;126(4):828-835.e3. doi: 10.1016/j.jaci.2010.06.049. PMID 20810155
- [Derived] Rothenberg ME, Klion AD, Roufosse FE, Kahn JE, Weller PF, Simon HU, Schwartz LB, Rosenwasser LJ, Ring J, Griffin EF, Haig AE, Frewer PI, Parkin JM, Gleich GJ; Mepolizumab HES Study Group. Treatment of patients with the hypereosinophilic syndrome with mepolizumab. N Engl J Med. 2008 Mar 20;358(12):1215-28. doi: 10.1056/NEJMoa070812. Epub 2008 Mar 16. PMID 18344568